CLINICAL TRIAL: NCT06283537
Title: The Effect of Online Episiotomy Simulation Training on Midwifery Students' Episiotomy Skill Performances, Satisfaction With the Teaching Method and Self-Confidence
Brief Title: Online Episiotomy Simulation Training for Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Nihal Aydin, Assistant Professor, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KÜBAP-01/2023-39
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Training Group, Sensitivity
Keywords: Episiotomy; Online Education; Simulation; Midwifery
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: A comparative randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: After all students in the face-to-face education and online education groups complete their applications, the students will practice on the material one by one in the school environment and will be evaluated through the Episiotomy Skill Evaluation Form. In the evaluation, a blinding technique will be used to prevent the person conducting the study interventions from making an evaluation in favor of the intervention group. For this purpose, the faculty member conducting the research initiatives will not take part in the evaluation, instead the evaluation will be made by two different field experts. The experts to be consulted for the evaluation will consist of people working as academicians in the field of obstetrics, nursing and midwifery. After the evaluation, students will have to fill out the survey (Student Information Form) and scale (Student Satisfaction and Self-Confidence in Learning Scale).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online episiotomy group (Experimental): 30 students will be assigned to the online education group with a random sampling model. To this group; Online episiotomy simulation training will be provided.
  Interventions: Other: Effect of training method
- Face to face training group (Experimental): 30 students will be assigned to the face-to-face education group with a random sampling model. This group will be given face-to-face episiotomy simulation training in the school environment, which is traditionally applied to the face-to-face training group..
  Interventions: Other: Effect of training method

INTERVENTIONS:
Other: Effect of training method — The effect of the training method given to midwifery students on their episiotomy application skills, satisfaction with the teaching method and self-confidence.

SUMMARY:
Purpose: To determine the effect of online episiotomy simulation training to midwifery students on their episiotomy application skills, satisfaction with the teaching method and self-confidence.

Method: This study is a randomized controlled experimental study. It will be conducted with third-year students studying at Kastamonu University Midwifery Department in the 2023-2024 period. In the research, all third-year students in the midwifery department (n=60) will be divided into 30 students into the online education group and 30 students into the face-to-face education group using a random sampling model. "Student Information Form", "Episiotomy Skill Evaluation Form" and "Student Satisfaction and Self-Confidence in Learning Scale" will be used to collect data.

DETAILED DESCRIPTION:
Episiotomy is the most commonly performed obstetric surgical procedure in obstetrics clinics. Failure to perform the procedure correctly may cause psychological and physiological problems in women. It is of great importance that midwives who are responsible for this practice receive training to acquire the necessary knowledge and skills. Midwifery students are expected to have sufficient skills in episiotomy practice before graduation. Teaching episiotomy practice is one of the basic skills taught face-to-face with simulation support. However, with the emergency distance education system implemented due to sudden decisions made in education and training after extraordinary situations such as pandemics and earthquakes, many theoretical and skill trainings had to be done online. It is not possible to predict whether similar extraordinary situations will occur again in the future. For this reason, it is considered important to evaluate the effect of online training on an important skill such as episiotomy application on students' episiotomy performance skills and their satisfaction with this training method and their self-confidence.

This study will be conducted to determine the effect of online episiotomy simulation training to midwifery students on their episiotomy application skills, satisfaction with the teaching method and self-confidence.

This study is a randomized controlled experimental study. It will be conducted with third-year students studying at Kastamonu University Midwifery Department in the 2023-2024 period. In the study, all 3rd year midwifery undergraduate students (n=60) taking the Normal Birth and Post-Care course will be included. 30 students will be allocated to the online education group and 30 students to the face-to-face education group using a random sampling model. To the online education group; Online episiotomy simulation training will be provided, while the face-to-face training group will be given face-to-face episiotomy simulation training in the traditionally applied school environment.

After all students in the face-to-face education and online education groups complete their applications, the students will practice on the material one by one in the school environment and will be evaluated through the Episiotomy Skill Evaluation Form. In the evaluation, a blinding technique will be used to prevent the person conducting the study interventions from making an evaluation in favor of the intervention group. For this purpose, the faculty member conducting the research initiatives will not take part in the evaluation, instead the evaluation will be made by two different field experts. The experts to be consulted for the evaluation will consist of people working as academicians in the field of obstetrics, nursing and midwifery. After the evaluation, students will have to fill out the survey (Student Information Form) and scale (Student Satisfaction and Self-Confidence in Learning Scale).

ELIGIBILITY:
Inclusion Criteria:

* Wanting to participate in the study voluntarily
* Having taken the normal birth and postpartum period course
* Not having any previous episiotomy experience

Exclusion Criteria:

* Student wants to leave the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
episiotomy skill performances | 4 weeks
  Is there a difference in episiotomy skill performance between midwifery students receiving online episiotomy simulation training and face-to-face episiotomy simulation training?Episiotomy skill performances will be evaluated with the "Episiotomy Skill Evaluation Form". Possible scores range from 0 to 100, with higher scores indicating higher performance for episiotomy skills. High scores indicate "high skill performance" and low scores indicate "low skill performance."

SECONDARY OUTCOMES:
Satisfaction with education | 4 weeks
  What is the satisfaction of midwifery students who receive episiotomy simulation training and face-to-face episiotomy simulation training? "Student Satisfaction and Self-Confidence in Learning scale" will be used in the evaluation. The minimum score obtained from the scale is 17 and the highest score is 61. A high score indicates high satisfaction and self-confidence.

OTHER OUTCOMES:
Self-confidence in learning | 4 weeks
  What is the learning self-confidence of midwifery students who receive episiotomy simulation training and face-to-face episiotomy simulation training? "Student Satisfaction and Self-Confidence in Learning scale" will be used in the evaluation. The minimum score obtained from the scale is 17 and the highest score is 61. A high score indicates high satisfaction and self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No